CLINICAL TRIAL: NCT02354846
Title: An Observational Study on Evaluating the Efficacy and Safety of Preemptive Antiviral Therapy With Tenofovir in HBsAg-positive Patients With Diffuse Large B-cell Lymphoma Receiving Rituximab-CHOP Chemotherapy (SPEED Study)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2014-0928
Record Dates: First submitted 2015-01-11; First posted 2015-02-03 (Estimated); Last update posted 2018-07-17 (Actual); Status verified 2018-07

CONDITIONS: B-cell Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
An Observational Study on Evaluating the Efficacy and Safety of Preemptive Antiviral Therapy with Tenofovir in HBsAg-positive Patients with Diffuse Large B-cell Lymphoma Receiving Rituximab-CHOP Chemotherapy (SPEED study)

ELIGIBILITY:
Inclusion Criteria:

* Males or females aged more than18
* HBsAg-positive DLBCL patients (it is possible to enrol the patients with combined DLBCL and low grade lymphoma such as follicular lymphoma)
* Previously untreated DLBCL patients who are suitable for receiving R-CHOP chemotherapy
* Serum ALT no more than 2 x ULN (including normal ALT)
* Life expectancy 6 months
* A negative serum or urine pregnancy test prior to treatment must be available both for pre menopausal women and for women who are no more than 1 years after the onset of menopause.
* Informed consent

Exclusion Criteria:

* Other subtype of lymphoma except DLBCL
* DLBCL patients who are NOT suitable for receiving R-CHOP chemotherapy OR plan to receive other chemotherapy
* patients had been treated with antiviral therapy known to have activity against HBV (e.g., alpha-interferon, lamivudine, telbivudine, clevudine, adefovir, entecavir or tenofovir) within the previous 6 months.
* evidence of hepatocellular carcinoma.
* evidence of decompensated liver disease

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Previously untreated Diffuse Large B-cell Lymphoma (DLBCL) with HBsAg (+) who are suitable for receiving R-CHOP chemotherapy
Sampling Method: Non-Probability Sample
Enrollment: 112 (Estimated)
Dates: Start 2015-02 (Actual); Primary Completion 2021-03 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
Percentage number of patients with hepatitis due to HBV reactivation | 2 years (every 3 months)
  Percentage number of patients with hepatitis due to HBV reactivation during the preemptive tenofovir therapy and for 24 weeks after withdrawal from tenofovir.
  Definition;
  * Hepatitis was defined as a more than 3-fold increase of serum ALT on 2 consecutive determinations at least 5 days apart.
  * Hepatitis was defined to be due to HBV reactivation when it was preceded or accompanied by an increase of serum HBV DNA to more than 10 times that of the pre-exacerbation baseline and the serum HBV DNA turned from negative to positive.
Percentage number of patients with hepatitis due to Safety assessment | 2 years (every 3 months)
  Safety assessment; NCI CTCAE v 4.0 and tolerability evaluation - drug compliance
Chemotherapy disruption due to hepatitis | 2 years (every 3 months)
  Chemotherapy disruption due to hepatitis: defined as either premature termination or delay of more than 8 days between chemotherapy cycles.

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Kim DY, Kim YR, Suh C, Yoon DH, Yang DH, Park Y, Eom HS, Lee JO, Kwak JY, Kang HJ, Hyun SY, Jo JC, Chang MH, Yoo KH, Lim SN, Shin HJ, Kim WS, Kim IH, Kim MK, Kim HJ, Lee WS, Mun YC, Kim JS. A Prospective Study of Preemptive Tenofovir Disoproxil Fumarate Therapy in HBsAg-Positive Patients With Diffuse Large B-Cell Lymphoma Receiving Rituximab Plus Cyclophosphamide, Doxorubicin, Vincristine, and Prednisone. Am J Gastroenterol. 2023 Aug 1;118(8):1373-1380. doi: 10.14309/ajg.0000000000002185. Epub 2023 Jan 13. PMID 36728217